CLINICAL TRIAL: NCT01812421
Title: A Nested Case-control Study on the Secondary Prevention of Ischemic Stroke and TIA by Hypertension Health Education Protocol (HHEP): The Post-Stroke Preventive Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Prevention
Other Study IDs: B2013-036-01
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: To Investigate the Relationship Between the Adherence of HHEP After ISTIA and Stroke Recurrence or Cardiovascular Events.

ARMS (1):
- Ischemic Stroke or TIA (ISTIA) patients (Experimental)
  Interventions: Other: Hypertension Health Education Protocol (HHEP)

INTERVENTIONS:
Other: Hypertension Health Education Protocol (HHEP)

SUMMARY:
Patients with a diagnosis of ischemic stroke or TIA (ISTIA), who are treated at hospital are asked to participate in our pre specified hypertension health education protocol (HHEP) after discharge from our hospital.HHEP was used as secondary prevention treatments of stroke and cardiovascular diseases.

HHEP consists of several items such as controlling the patient's hypertension level, monitoring the adherece of antihypertensive agents, reducing risk factors of hytertension like tobacco smoking, obesity, and motivating the patient to physical activity and to a healthy diet.

Patients will receive visits by a study nurse with the aim of supervising, monitoring, and recording the adherence of HHEP. The patients will be classified as different adherence level at the end of the study according to their adherence condition.

This study is aimed at testing the hypothesis that controlling hypertension and its risk factors was more effective than those do not receive HHEP in reducing the recurrence of stroke and cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

Participants were eligible for this observational cohort study if they were age 18 years or older; Hospitalized for a primary diagnosis of acute ischemic stroke or Transient Ischemic Attack (TIA) and concurrently diagnosed as hypertension; Provided consent to participate, and their data can be collected from Medical Record System of our hospital.

Exclusion Criteria:

We will exclude people who are onset of symptoms 3 months after their ischemic stroke or TIA; The stroke events occurred before the baseline survey were identified from the Hospital Discharge Register retrospectively and excluded from the analyses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Nonfatal vascular events: ischemic or hemorrhagic stroke recurrence (ICD-9 431 or ICD-10 I61), or myocardial infarction(MI) (ICD-9 410 or ICD-10 I21). | 1 year

SECONDARY OUTCOMES:
vascular death (death within 30 days after a vascular event) and all-cause mortality. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Brain Center,Guangdong Province Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong, China